CLINICAL TRIAL: NCT00774007
Title: Effect of Mesalazine on Low Grade Mucosal Inflammation in Irritable Bowel Syndrome. A Pilot Double Blind Placebo Controlled Study.
Brief Title: A Randomized Controlled Pilot Trial of Mesalazine in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: SOFAR S.p.A. (Industry)
Collaborators: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Dr. Giovanni Barbara, Department of Internal Medicine and Gastroenterology, University of Bologna, Bologna, ITALY
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IBS-01/03
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome, abdominal pain, abdominal bloating, immune cells, mast cells
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- Mesalazine (Active Comparator): mesalazine 800 mg t.i.d.
  Interventions: Drug: mesalazine

INTERVENTIONS:
Drug: mesalazine
  Arms: Mesalazine
Drug: placebo
  Arms: Placebo

SUMMARY:
Emerging evidence indicates the presence of low-grade mucosal inflammation and its pathogenetic role in IBS. The aim of this pilot study is to provide that mesalazine treatment of IBS patients reduces low grade colonic inflammation.

DETAILED DESCRIPTION:
Emerging evidence indicates the presence of low-grade mucosal inflammation and its pathogenetic role in IBS. The aim of this pilot study is to provide that mesalazine treatment of IBS patients reduces low grade colonic inflammation.

This is a pilot double blind placebo controlled study.

A total of twenty patients (both males and females) will be recruited; ten will be randomly assigned to the placebo controlled arm and ten to the study medication arm.

Inclusion criteria:

* IBS patients (both males and females) with positive diagnosis based on Rome II criteria [20]
* age ≥ 18 years
* Patients capable of conforming to the study protocol;
* Patients who have given their free and informed consent

Exclusion criteria:

- Patients with ascertained Inflammatory Bowel Diseases (Crohn disease, Diverticular disease, Ulcerative colitis, Infectious colitis, Ischemic colitis, microscopic colitis); food intolerance/allergy; active malignancy of any type, or history of a malignancy; presence of major abdominal surgeries; ascertained hypersensitivity to the salicylates; positive faecal culture for bacterial, mycotic or parasitic pathogens; patients with history of clinically significant renal (creatinine ≥ 2.0 mg/dL or ≥177 μmol/L), hepatic (AST or ALT greater than three times the upper limit of normal range), cardiac, metabolic or haematological disease; esophageal, gastric or duodenal ulcer within 30 days prior to randomization; patients with intended or ascertained pregnancy; lactation; patients who become unable to conform to protocol; patients who are continuously taking laxatives; patients in antibiotic therapy during the last month; patients in current therapy with corticosteroids; treatment with any investigational drug within the previous 30 days; treatment with lactulose or with any compound that lowering the colonic pH can prevent the release of the active moiety; recent history or suspicion of alcohol abuse or drug addiction; any severe pathology that can interfere with the treatment or the clinical tests of the trial; previous participation in this study.

Treatments:

Mesalazine cpr 800 mg t.i.d. for 8 weeks Placebo cpr t.i.d. for 8 weeks

Primary End Points:

The primary end point of the study will be to assess the effect of mesalazine treatment on:

• Total number of inflammatory mucosal cells

Secondary End Points:

* Individual inflammatory cell subsets and enterochromaffin (EC) cells in the colonic mucosa (mast cells, macrophages, B and T lymphocytes subsets)
* Inflammatory release by mucosal biopsies
* Indicative measures of symptoms relief

The local tolerability of treatment, through the daily monitoring of intolerance manifestations at the gastrointestinal level, will be carried out by each patient and reported to the investigator on each control visit.

Adverse event(s) and concurrent illness(es) which occur during the study will be monitored.

The following laboratory test results will be recorded at Basal Visit (T0) and at the end of the study (T8):

• Hemochrome, AST , ALT, creatinine, γ-GT, alkaline phosphatase (AP), total bilirubin, glucose, N, Na+, K+, Ca 2+ Urine pregnancy test: if the patient is a female of childbearing potential, a urine pregnancy test will be performed and must be confirmed as negative before the first dose of study medication is administered.

On the BASAL VISIT (T0) the following will be performed:

1. Diagnosis of IBS disease based on Rome II criteria
2. Check inclusion and exclusion criteria
3. Written Consent
4. Record medical history and concomitant medication
5. Physical examination
6. Urine pregnancy test
7. Vital Signs (BP, HR, LR)
8. Fecal Culture
9. Sigmoid biopsy
10. Delivery of the patient's diary
11. Laboratory Assessments
12. Symptom questionnaire

On the VISITS T2, T4 and T6 ( after 2, 4 and 6 weeks) the following will be performed:

1. Symptom questionnaire
2. Vital Signs (BP, HR, LR)
3. Collection/Delivery of the patient's diary
4. Record Adverse Events
5. Record Concomitant Medication

On the VISIT T8 or FINAL VISIT (After eight weeks) the following will be performed:

1. Sigmoid biopsy
2. Symptom questionnaire
3. Collection/Delivery of the patient's diary
4. Physical examination
5. Laboratory Assessments
6. Vital Signs (BP, HR, LR)
7. Record Adverse Events
8. Record Concomitant Medication Data recorded during the study will be summarised by treatment group and compared using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* IBS patients (both males and females) with positive diagnosis based on Rome II criteria
* age ≥ 18 years
* Patients capable of conforming to the study protocol;
* Patients who have given their free and informed consent

Exclusion Criteria:

* Patients with ascertained Inflammatory Bowel Diseases (Crohn disease, Diverticular disease, Ulcerative colitis, Infectious colitis, Ischemic colitis, microscopic colitis)
* Patients with ascertained food intolerance/allergy
* Patients with active malignancy of any type, or history of a malignancy (patients with a history of other malignancies that have been surgically removed and who have no evidence of recurrence for at least five years before study enrollment are also acceptable)
* Presence of major abdominal surgeries
* Ascertained hypersensitivity to the salicylates
* Positive faecal culture for bacterial, or parasitic pathogens
* Patients with history of clinically significant renal (creatinine ≥ 2.0 mg/dL or ≥177 μmol/L), hepatic (AST or ALT greater than three times the upper limit of normal range), cardiac, metabolic or haematological disease
* Esophageal, gastric or duodenal ulcer within 30 days prior to randomization
* Patients with intended or ascertained pregnancy; lactation
* Patients who become unable to conform to protocol
* Patients who are continuously taking laxatives
* Patients in antibiotic therapy during the last month
* Patients in current therapy with corticosteroids
* Treatment with any investigational drug within the previous 30 days
* Treatment with lactulose or with any compound that lowering the colonic pH can prevent the release of the active moiety
* Recent history or suspicion of alcohol abuse or drug addiction
* Any severe pathology that can interfere with the treatment or the clinical tests of the trial
* Previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in the study was to assess the effect of mesalazine treatment on total number of mucosal immune cells in the colonic mucosa of patients with IBS. | 8 weeks

SECONDARY OUTCOMES:
Effect of mesalazine on: 1) mucosal immune cell subsets; 2) inflammatory mediator release from mucosal biopsies; 3) symptom relief, as detected by means of visual analogue scales. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Barbara, MD, Principal Investigator — University of Bologna; Roberto Corinaldesi, MD, Study Chair — University of Bologna
Locations (1):
- Department of Internal Medicine & Gastroenterology, Bologna, Italy